CLINICAL TRIAL: NCT02160769
Title: The Assessment of Tear Layer and Tear Layer Lipid Distribution Pre and 1 Month Post Pterygium Surgery Using a LipiView Ocular Surface Interferometer (LipiView)
Brief Title: Tear Layer Lipid Thickness in Pterygium Patient Before and After Surgery
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Other Study IDs: R1075/90/2013; 2013/851/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Dry Eye
Keywords: Tear Lipid Thickness; Pterygium surgery
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators study aims to capture the objective effects of pterygium surgery on tear layer lipid thickness and the tear layer.

Previous objective studies of the tear film has been limited to corneal staining grading, tear break up time and Schirmer's test which have been shown to poor to moderate repeatability. The effect of pterygiums on tear layer lipid thickness (LLT) has not previously been explored. With the LipiView Ocular Surface Interferometer, the investigators have the ability to assess the optical coherence interference pattern produced by light reflected off the tear film in a safe and non-invasive manner. Software analysis of the image then measures the tear LLT which can be used to objectively quantify the diagnosis of lipid-deficient dry eye.

DETAILED DESCRIPTION:
Pterygium is a condition characterized by abnormal conjunctival growth on the cornea and is particularly prevalent in tropical climates. In severe circumstances, it may lead to visual loss by obscuration of the visual axis and inducing corneal astigmatism (1). It is often also associated with dry eye symptoms and studies have previously shown some correlation with shortened tear break up time (TBUT)(2) but not Schirmer's Test (3).

Schirmer's Test, corneal staining and TBUT are often used to investigate symptoms of dry eyes but the diagnosis and assessment is often difficult due to the poor repeatability of the tests(4). Treatments for dry eyes often rely on patient's subjective symptomatic improvements as a measure of outcome although no literature has been published of subjective symptoms for pterygium patients. The effects of pterygium surgery and tear lipid layer thickness has also not been studied.

The LipiView Ocular Surface Interferometer is a HSA-approved imaging device that allows clinicians evaluate the characteristics and thickness of the tear lipid layer thickness (LLT) in a safe and non-invasive manner. The device utilizes white light from a LED source that is directed at the tear film over the inferior corneal region. Reflected light is captured by a high resolution camera and the optical inference pattern is evaluated by software to determine the LLT (5). It also was found to correlate with other dry eye diagnostic tests, such as tear film break-up time (TBUT), Schirmer's test and corneal staining(6,7). LLT is also reported to better correlate with symptoms than other objective dry eye tests(5).

LipiView was also capable of detecting a significant change in longitudinal lipid thickness in 10 patients one month after blepharoplasty. A similar result may be obtained from the investigators patients post pterygium surgery.

This current study aims to investigate the effects of pterygium surgery on tear lipid layer thickness with LipiView. The results will be compared with the effects of pterygium surgery on TBUT, and corneal staining. The subjective improvement in dry eye symptoms post pterygium surgery will also be studied.

Clinical importance This study can provide further data to support pterygium surgery as a role in dry eyes management in an objective and reproducible manner. New data on pterygium and tear lipid layer thickness as well as subjective dry eye symptoms will also be explored.

Study Objectives and Purpose The Assesssment of Dry Eye Symptoms, Tear Layer and Tear Layer Lipid Thickness Pre and 1month Post Pterygium Surgery using a LipiView Ocular Surface Interferometer (LipiView)

Study design:

Prospective study

Rationale:

Methods:

Participants and target sample size Target sample size: 80 40 patients who will be undergoing pterygium surgery will be recruited for this study. Another 40 patients will be recruited from the general ophthalmology (ECS) clinic. These patients are cleared to have no lid disturbances in terms of function or anatomy, and will serve as the "control" group.

Permission will be sought from the junior ophthalmologists and the supervising ophthalmologist (in the event of a training list) or from the senior ophthalmologist if he is performing the surgery himself. These patients would have been diagnosed with pterygium and opted for surgical excision and conjunctival autograft. Pre operatively they will complete a simple questionnaire to evaluate any dry eye symptoms. Participants will be examined under the slit lamp for fluorescein dye corneal staining and fluorescein dye tear break up time. The patients will then undergo a LipiView Ocular Surface Interferometer Measurement of Tear lipid layer thickness.

Visit schedules Two/Three visits is required for paticipants who are undergoing pterygium surgery.

Only one visit is required for normal controls who are recruited from general ophthalmology (ECS) clinic.

Duration of study:

10 months.

Procedures:

1. Assessment of Dry Eye Symptoms (SANDE) Participants will be asked to score and fill up a dry eye questionnaire that assesses the symptomatic severity and frequency of dry eyes symptoms.

   • SANDE Questionnaire Consists of 3 questions on frequency and severity. VAS will be applied to evaluate dry eye symptoms as described by Schaumberg et al. (Schaumberg, Gulati et al. 2007). The scores will be recorded separately for frequency and severity of dry eye symptoms. Patients will be asked to mark "X" on a 100mm line that corresponds to the degree of the symptom. A global score will be calculated by multiplying the frequency score by the severity score and taking the square root of the result (to transform back to the original scale).

   Basic biodata such as age, race, gender will also be recorded.
2. LipiView Ocular Surface Interferometer Measurement of Tear lipid Layer Thickness

   Prior measuring the tear lipid layer thickness, participants are advised not to:

   i. instill any eye ointment for at least 24 hours, or ii. instill eye drops or wear contact lenses for 4 hours, or iii. swim in a chlorinated pool, rub their eyes or put on eye cosmetics on the day of the measurement.

   During the measurement of each eye, the participants place their chins on a chin rest and look at a single white light source for 30 seconds. During this period, participants are encouraged to blink freely at a comfortable rate which the assessor measures the LLT.

   Similar steps would be taken for the other eye as a control eye.

   Assessment of fluorescein tear break up time and corneal staining will be conducted only after LipiView LLT measurement.
3. Fluorescein Dye Tear Break-up Time (TBUT) Fluorescein dye is introduced onto the lower eyelid by a wetted fluorescein strip. The tear film will then be observed with blue light using a slit lamp to the point where it breaks. The time from the previous blink to the breaking of the tear film will be recorded to the nearest second.
4. Fluorescein Dye Corneal Staining After fluorescein dye is introduced, the cornea will be examined for green stains indicating epithelial erosion, a sign of damage due to dryness. The number of green stains and their location on the cornea (superior, central, inferior, temporal, nasal fields) will be recorded.
5. Patient will undergo pterygium excision and conjunctival autograft on the prearranged surgery date.
6. Steps 1-4 will be repeated 1 month post operatively.

Outcomes:

Primary outcome:

An increase in tear lipid layer thickness 1 month post pterygium surgery in the operated eye.

Statistics:

There will be no interim analysis. Analysis will be performed after all the subjects have completed the required visits or have withdrawn from the study.

Data will be analysed for sample mean of pre and post-operative questionnaire score, tear break up time, corneal staining and tear lipid layer thickness in both the operated and un-operated eye. The confidence intervals of the pre and post-operative in both the operated and un-operated will be calculated with T-test analysis.

Expected outcomes:

There should be decreased dry eye symptoms in the operated pterygium eye with a improvement in tear break up time, decreased corneal staining and increase tear lipid layer thickness when compared to pre operative.

Potential problems No potential problems are expected for this study.

Inclusion Criteria

1. Normal controls or patients with pterygium who have consented for pterygium surgery and are willing to participate in this study

Exclusion Criteria

1. Active ocular surface conditions such as infections.
2. Any other specified reason as determined by clinical investigator.

ELIGIBILITY:
Inclusion Criteria:

* Normal controls or patients with pterygium who have consented for pterygium surgery and are willing to participate in this study

Exclusion Criteria:

* Active ocular surface conditions such as infections.
* Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normal volunteers and Pterygium patients undergoing surgery to remove Pterygium
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
tear lipid layer thickness | 1 month
  An increase in tear lipid layer thickness 1 month post pterygium surgery in the operated eye

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore., Singapore